CLINICAL TRIAL: NCT06259253
Title: Understanding Patient Experience Among Asians at MD Anderson
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0521; NCI-2024-00901 (Registry Identifier: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-01-30; First posted 2024-02-14 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Cohort 1 - Patient/Provider: Participant will complete a computer-based questionnaire about your age, gender, income, highest level of education, patient experience, medical mistrust, social support and health care access.
- Observational Cohort 2 - Patient/Provider: Participant will complete a computer-based questionnaire about your age, gender, income, highest level of education, patient experience, medical mistrust, social support and health care access.

SUMMARY:
The purpose of this research study is to understand barriers to and facilitators of a positive patient experience for Asian patients.

DETAILED DESCRIPTION:
Primary Objective:

a. Identify critical aspects of inpatient experience among former Asian/Asian American patients at MD Anderson.

Secondary Objectives:

a. Determine MD Anderson health care providers' perceptions of Asian/Asian American inpatient experience.

ELIGIBILITY:
Inclusion criteria for former patients:

* Self-identify as Asian/Asian American
* Are 18 years or older
* Have been diagnosed with cancer, any type
* Received inpatient care at MD Anderson between 2019 and 2022
* Have a U.S. address
* Can read and write in English or simplified Chinese

Exclusion criteria for former patients:

• None

Inclusion criteria for healthcare providers:

* Self-report as a practicing inpatient provider (advanced practice provider, hospitalist, physician, nurse) at MD Anderson
* Treated patients diagnosed with breast, colon, prostate, thyroid, or lymphatic cancer
* Provided treatment services to Asian/Asian American patients between 2019 and 2022

Exclusion criteria for healthcare providers:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center Participants
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Picker Patient Experience Questionnaire (PPE-15) | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, MPH,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org